CLINICAL TRIAL: NCT02241135
Title: Phase I Safety and Immunogenicity Trial of an Investigational RNActive® Rabies Vaccine (CV7201) in Healthy Adults
Brief Title: RNActive® Rabies Vaccine (CV7201) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CV-7201-102; 2013-002171-17 (EudraCT Number)
Record Dates: First submitted 2014-08-22; First posted 2014-09-16 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-05

CONDITIONS: Rabies
Keywords: Rav G protein; rabies; VNT; immunogenicity; PrEP vaccination; mRNA; CV7201
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 80 µg CV7201 mRNA short (Experimental): Vaccination by injection on days 0, 7, 28.
  Interventions: Biological: CV7201 mRNA
- 160µg CV7201 mRNA short (Experimental): Vaccination by injection on days 0, 7, 28.
  Interventions: Biological: CV7201 mRNA
- 80 µg CV7201 mRNA long (Experimental): Vaccination by injection on days 0, 28, 56.
  Interventions: Biological: CV7201 mRNA
- 160 µg CV7201 mRNA long (Experimental): Vaccination by injection on days 0, 28, 56.
  Interventions: Biological: CV7201 mRNA
- 320 µg CV7201 mRNA long (Experimental): Vaccination by injection on days 0, 28, 56.
  Interventions: Biological: CV7201 mRNA
- 640 µg CV7201 mRNA long (Experimental): Vaccination by injection on days 0, 28.
  Interventions: Biological: CV7201 mRNA
- 200 µg CV7201 mRNA long (Experimental): Vaccination by injection on days 0, 28, 56.
  Interventions: Biological: CV7201 mRNA
- 400 µg CV7201 mRNA long (Experimental): Vaccination by injection on days 0, 28, 56.
  Interventions: Biological: CV7201 mRNA

INTERVENTIONS:
Biological: CV7201 mRNA — CV7201 is composed of 1 RNActive® mRNA that encodes the rabies virus glycoprotein.
  Other Names: CV7201 messenger RNA; CV7201 RNActive®

SUMMARY:
The purpose of this trial is to assess the safety and immunogenicity of an investigational RNActive® rabies vaccine (CV7201) in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers aged 18 to 40 years inclusive
2. Compliant with protocol procedures and available for clinical follow-up through the last planned visit (V9)
3. Physical examination and laboratory results without clinically significant findings
4. Body Mass Index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2
5. Females: Negative human chorionic gonadotropin (HCG) pregnancy test (serum) for women presumed to be of reproductive potential on the day of enrolment
6. Females of childbearing potential must use acceptable methods of birth control during the trial and Follow-up period (from 6 weeks before the first administration of the test vaccine for the duration of the trial i.e., until the last planned visit (V9)). The following methods of birth control are acceptable when used consistently and correctly: established use of oral, injected or implanted hormonal methods of contraception; intrauterine devices (IUDs) or intrauterine systems (IUSs) with the exception of steel or copper wire; barrier methods of contraception (condom or occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository); true abstinence (periodic abstinence [e.g., calendar, ovulation, symptothermal and postovulation methods] and withdrawal are not acceptable).
7. Males must use reliable forms of contraception (barrier method with spermicidal agent or true abstinence) and must refrain from sperm donation during the trial and Follow-up period i.e., until the last planned visit (V9).

Exclusion Criteria:

1. Use of any investigational or non-registered product (drug or vaccine) other than the trial vaccine within 4 weeks preceding the administration of the trial vaccine, or planned use during the trial period
2. Subject has received any other licensed vaccines within 4 weeks prior to the administration of the trial vaccine
3. Subject has received any investigational or licensed rabies vaccine previously
4. Intending to travel to regions/countries for which rabies vaccinations are recommended or where high risk of infections exists according to travel recommendations by the German Society of Tropical Medicine and International Health (DTG) during the trial and up to V9 (Day 91/120) Follow-up
5. Any treatment with immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the trial vaccine. The use of inhaled and nasal steroids, as well as topical steroids outside the vaccination area, will be permitted
6. Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination
7. History of autoimmune disease
8. Administration of immunoglobulins (Igs) and/or any blood products within the 3 months preceding the administration of the trial vaccine
9. Subject is taking chloroquine for malaria treatment or prophylaxis
10. Acute disease at the time of enrolment. Acute disease is defined as the presence of a moderate or severe illness or fever ≥ 38 °C measured orally
11. Presence or evidence of significant acute or chronic, uncontrolled medical or psychiatric illness (subjects with uncomplicated chronic diagnoses stable and treated for ≥ 3 months e.g., mild hypertension well-controlled with medication, may be enrolled - provided the condition and its therapy are known not to be associated with an immunocompromised state or an autoimmune disease
12. Major congenital defects
13. Known allergy to any component of the trial product i.e., protamine. This includes subjects with allergy to fish protein, diabetics with allergy to protamine-containing insulin, or post-vasectomy males
14. Known type I allergy to beta lactam antibiotics
15. Evidence of current alcohol or drug abuse
16. History of any neurological disorders or seizures, with the exception of febrile seizures during childhood
17. Seropositivity for human immunodeficiency virus (HIV), hepatitis B virus (HBV) (except in subjects previously vaccinated against HBV) or hepatitis C virus (HCV)
18. Foreseeable non-compliance with protocol as judged by the Investigator
19. For females: Pregnancy or lactation
20. History of any life-threatening anaphylactic reactions.
21. Subjects with impaired coagulation in whom an IM injection is contraindicated.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2013-10; Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of serious adverse events (SAEs)/adverse events (AEs) and local tolerability assessment of the vaccination site | up to 64 days after the last vaccination
  The occurrence of AEs will be assessed by non-directive questioning of the subject at each visit. Further, AEs volunteered by the subject during or between visits - as subject diary card entries - or detected through observation, physical examination, laboratory test, or other assessments during the entire observation period, will be documented. Subjects will be instructed that they must immediately report any AEs, subjective complaints or objective changes in their well-being to the Investigator or the clinic personnel, regardless of the perceived relationship between the event and the test product. The Investigator is responsible for reporting all AEs in the eCRF that are observed or described by the subject, regardless of their relationship to the trial vaccine or their clinical significance.

SECONDARY OUTCOMES:
The lowest CV7201 dose to elicit rabies VNTs ≥ 0.5 IE/ml | Rabies VNTs measured 14 days after the 3rd vaccination (Visit 8)
  Rabies virus neutralizing titers (VNTs) measured in serum blood samples taken 14 days after the the last vaccination (Visit 8).
Number of treatment discontinuation due to IMP-related AEs/SAEs | up to 64 days after the last vaccination
  Number of subjects discontinued from treatment after the first or second vaccination due to vaccination-related reactions or AEs/SAEs.
  Period for observation in order to decide on withdrawal of subjects from next vaccination starts with Visit 1 (day 0, first vaccination) and lasts until the day of the third scheduled vaccination (pre-vaccination examination).

CONTACTS AND LOCATIONS:
Overall Officials: Franz-Josef Falkner von Sonnenburg, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Abteilung für Infektions- und Tropenmedizin der Ludwig-Maximilians-Universität, Munich, Germany

REFERENCES:
- [Derived] Alberer M, Gnad-Vogt U, Hong HS, Mehr KT, Backert L, Finak G, Gottardo R, Bica MA, Garofano A, Koch SD, Fotin-Mleczek M, Hoerr I, Clemens R, von Sonnenburg F. Safety and immunogenicity of a mRNA rabies vaccine in healthy adults: an open-label, non-randomised, prospective, first-in-human phase 1 clinical trial. Lancet. 2017 Sep 23;390(10101):1511-1520. doi: 10.1016/S0140-6736(17)31665-3. Epub 2017 Jul 25. PMID 28754494